CLINICAL TRIAL: NCT02840955
Title: The Effect of Gladskin on Disease Severity and the Skin Microbiome, Including Staphylococcus Aureus, in Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Micreos (Unknown); TNO (Other); Regional Public Health Laboratory Kennemerland (Unknown)
Responsible Party: Principal Investigator, Suzanne G.M.A. Pasmans, Prof., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-233
Record Dates: First submitted 2016-07-11; First posted 2016-07-21 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Staphylococcus aureus; Microbiome; Staphefekt
MeSH Terms: conditions — Dermatitis, Atopic; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Staphefekt SA.100 (Active Comparator): Staphefekt SA.100 cream, twice daily on (lesional) skin during 12 weeks
  Interventions: Device: Staphefekt SA.100
- Placebo (Placebo Comparator): Placebo (Gladskin cream without the Staphefekt protein), twice daily on (lesional) skin during 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Staphefekt SA.100
  Other Names: Gladskin
  Arms: Staphefekt SA.100
Other: Placebo
  Arms: Placebo

SUMMARY:
Colonization with Staphylococcus aureus is related to inflammation in atopic dermatitis. Gladskin is a product for topical use containing the proprietary enzyme Staphefekt SA.100, which has the ability to specifically lyse the cell wall of S. aureus. The investigators hypothesize that Staphefekt decreases S. aureus colonization of the skin and consequently decreases symptoms of atopic dermatitis.The goal of this study is to determine the effect of Staphefekt on the use of topical corticosteroids in patients with atopic dermatitis. Secondary goals are to retrieve information about the effect on clinical symptoms, quality of life, growth characteristics of Staphylococcus aureus and the further microbiome.

DETAILED DESCRIPTION:
This is a multi center intervention study with a placebo controlled, double blind and randomized design. After standardization of corticosteroid treatment (triamcinolone acetonide 0.1% cream), patients will be randomized in a 1:1 fashion to either treatment with Staphefekt SA.100 for 12 weeks or treatment with a placebo for 12 weeks. Topical corticosteroid use will be evaluated 2, 6, 12 and 20 weeks after start of the intervention. Swabs of the skin, nose and throat will be collected at baseline, week 2, 12 and 20.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis of moderate and severe severity. Defined by EASI score of 7.1 to 50 performed by the researcher at visit 1
* Topical corticosteroid use (of any type)
* 18 years or older
* Able to read patient information and provide informed consent

Exclusion Criteria:

* Use of systemic antibiotics or corticosteroids in the previous 2 months
* Use of Methotrexate or oral immunosuppressive agents in the previous 3 months
* Use of topical antibiotics in the previous 7 days
* Use of light therapy in the previous 3 months
* Use of Gladskin in the previous 7 days
* Contact allergy to components of the study drug (e.g., propylene glycol and glycerol)
* Clinically infected atopic dermatitis
* Existence of another skin condition, such as folliculitis or psoriasis that could interfere with the assessment of the eczema severity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Difference in number of days/week corticosteroid use between verum and placebo group over 12 weeks | baseline, 12 weeks

SECONDARY OUTCOMES:
Difference in mean grams/week topical corticosteroid use between verum and placebo group | baseline, 12 and 20 weeks
Proportion of patients with AD who indicate to have used less corticosteroids at week 2 and 12, as compared to baseline and at week 20 as compared to the 12 week treatment period | baseline, 2, 12 and 20 weeks
Change in Eczema Area and Severity Index (EASI) from baseline to week 2, 6, 12 and 20 | baseline, 2, 6, 12 and 20 weeks
Change in Patient Orientated Eczema Measurement (POEM) from baseline to week 2, 6, 12 and 20 | baseline, 2, 6, 12 and 20 weeks
Change in Investigator Global Assessment (IGA) scale from baseline to week 2, 6 and 12 and week 20 | baseline, 2, 6, 12 and 20 weeks
Change in Pruritus Numerical Rating Scale (Pruritus NRS) from baseline to week 2, 6, 12 and week 20 | baseline, 2, 6, 12 and 20 weeks
Mean time to flare from baseline through week 12 and from week 12 through week 20. Flare is defined is an exacerbation that requires the need of any stronger topical therapy, an increase in dosage of the topical therapy or the need of a systemic therapy. | baseline, 12 and 20 weeks
Number of flares through week 12 | baseline, 12 weeks
Change in Skindex-29 score from baseline to week 12 and week 20 | baseline, 12 and 20 weeks
Proportion of patients with a reduction of S. aureus from baseline to measurement 1 (0,5 hour after baseline) as determined by semi quantitative culture | baseline, 1 day
Proportion of patient with a > 1 log reduction of S. aureus from the lowest measurement (visit 1 or visit 2a) to week 2 and week 12 as determined by quantitative polymerase chain reaction (qPCR) | baseline (visit 1 or 2a), 2 and 12 weeks
Change in relative abundance of bacteria: determined by 16 Svedberg units ribosomal ribonucleic acid (16s rRNA) sequencing | baseline, 2, 12 and 20 weeks
Incidence of (serious) adverse device events from baseline through the end of the study, evaluated by medical check-ups, including vital signs | baseline, 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Centre, Rotterdam, Netherlands

REFERENCES:
- [Derived] Totte J, de Wit J, Pardo L, Schuren F, van Doorn M, Pasmans S. Targeted anti-staphylococcal therapy with endolysins in atopic dermatitis and the effect on steroid use, disease severity and the microbiome: study protocol for a randomized controlled trial (MAAS trial). Trials. 2017 Aug 31;18(1):404. doi: 10.1186/s13063-017-2118-x. PMID 28859690